CLINICAL TRIAL: NCT01135329
Title: Reduced-intensity, Related-donor Allogeneic BMT With Fludarabine, Busulfan, and High-dose Posttransplantation Cyclophosphamide for Hematologic Malignancies
Brief Title: Reduced-intensity, Related-donor Bone Marrow Transplantation Followed by High-dose Cyclophosphamide for Hematologic Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The stopping rule was met and hence the study was closed
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1046; NA_00039363 (Other: JHM IRB)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Lymphoma; Leukemia; Myelodysplastic Syndrome
Keywords: Lymphoma; Hodgkin's lymphoma; Non hodgkin's lymphoma; Leukemia; Acute myeloid leukemia (AML); Acute lymphoblastic leukemia(ALL); Chronic myeloid leukemia (CML); Chronic Myelomonocytic (CMML); Myelodysplastic syndrome (MDS); High-risk acute leukemia in first remission; Relapsed leukemia in remission; Cyclophosphamide; High-dose cyclophosphamide; Fludarabine; Busulfan; Allogeneic; Nonmyeloablative; Reduced intensity; Haploidentical; Bone marrow transplant (BMT)
MeSH Terms: conditions — Lymphoma; Leukemia; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — fludarabine; fludarabine phosphate; Influenza Vaccines; Busulfan; Cyclophosphamide; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant (Experimental): Reduced-intensity transplant with a fludarabine- and busulfan-based preparative regimen. GVHD prophylaxis with cyclophosphamide, tacrolimus, and mycophenolate mofetil.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m^2 IV daily on Day -6 through Day -2.
  Other Names: Fludara; Flu
Drug: Busulfan — 1 mg/kg PO OR 0.8 mg/kg IV four times daily on Day -6 through Day -3.
  Other Names: Busulfex; Myleran
Drug: Cyclophosphamide — 50 mg/kg IV daily on Day +3 and Day +4.
  Other Names: CTX; Cytoxan; Cy
Drug: Mycophenolate Mofetil — 15 mg/kg PO three times daily (max daily dose of 3g) starting on Day +5.
  Other Names: MMF; CellCept
Drug: Tacrolimus — Dosed based on drug levels; begin on Day +5 at 1 mg IV daily.
  Other Names: FK506; FK-506; Prograf

SUMMARY:
This research is being done to learn more about reduced-intensity bone marrow transplantation (BMT), also known as a "mini" transplant for patients with blood cancers, using bone marrow from a relative.

The main goal of the study is to determine how quickly the donor's bone marrow "takes" in your body. Other goals include describing how many people accept the bone marrow and how quickly the blood counts come up; describing Graft-versus-host disease (GVHD) and other complications; and describing how many people survive without progressive cancer and survive overall

DETAILED DESCRIPTION:
At the present time there are few or no cures for people with cancer of the blood or lymph glands outside of a bone marrow transplant (BMT). BMT has developed over several decades of research as an effective treatment of various malignant and nonmalignant hematologic diseases.

This research is being done to learn more about reduced-intensity bone marrow transplantation (BMT), also known as a "mini" transplant for patients with blood cancers, using bone marrow from a relative. The bone marrow for this transplant comes from a relative who is a half-match or "haplo" match to you. Possible donors include parents, siblings, and children.

"Mini" transplants have been given to many people with various cancers but are considered experimental. Over 200 people at Johns Hopkins have received mini transplants with high doses of cyclophosphamide after the transplant. However, the chemotherapy combination and other treatment given before those transplants were different from what is in this study. Although all of the chemotherapy and immune-lowering drugs used in this study are approved by the Food and Drug Administration (FDA), the combination of medications used in this study are not FDA approved and are experimental.

ELIGIBILITY:
Inclusion Criteria:

* First-degree related donor who is at minimum HLA haploidentical
* Eligible diagnoses:

  1. Low-grade non-Hodgkin's lymphoma or plasma cell neoplasm that has progressed during multiagent therapy, failed at least two prior therapies (excluding single agent rituximab and single agent steroids), or in the case of lymphoma undergone histological conversion:

     * Follicular grade 1 or 2 lymphoma
     * Follicular lymphoma not otherwise specified
     * Marginal zone (or MALT) lymphoma
     * Lymphoplasmacytic lymphoma / Waldenstrom's macroglobulinemia
     * Hairy cell leukemia
     * Small lymphocytic lymphoma (SLL) or chronic lymphocytic leukemia (CLL)
     * Prolymphocytic leukemia
     * Low grade B-cell lymphoma, unspecified
     * Multiple myeloma
     * Plasma cell leukemia
  2. Poor-risk SLL or CLL, defined by an 11q or 17p deletion, histological conversion, or disease progression < 6 months after a purine analog-containing regimen
  3. Aggressive lymphoma that has failed at least one prior regimen of multiagent chemotherapy, and patient is either ineligible for autologous BMT or autologous BMT is not recommended:

     * Hodgkin lymphoma
     * Follicular grade 3 lymphoma
     * Mantle cell lymphoma or leukemia
     * Diffuse large B-cell lymphoma (excluding primary CNS lymphoma). Eligible subtypes include primary mediastinal large B-cell lymphoma, T-cell rich large B-cell lymphoma, and large B-cell lymphoma not otherwise specified.
     * Burkitt's lymphoma/leukemia
     * Atypical Burkitt's lymphoma/leukemia (high grade B-cell lymphoma, unclassified, including that with features intermediate between Burkitt's and diffuse large B-cell lymphoma)
     * Anaplastic large cell lymphoma
     * Plasmablastic lymphoma
     * Peripheral T-cell lymphoma
  4. Relapsed or refractory acute leukemia in second or subsequent remission
  5. Poor-risk acute leukemia in first remission
  6. AML with at least one of the following:

     * AML arising from MDS or a myeloproliferative disorder, or secondary AML
     * Presence of Flt3 internal tandem duplications
     * Poor-risk cytogenetics
     * Primary refractory disease

       * ALL (leukemia and/or lymphoma) with at least one of the following:
     * Adverse cytogenetics
     * Clear evidence of hypodiploidy
     * Primary refractory disease

       * Biphenotypic leukemia
       * MDS with at least one of the following features:
       * Poor-risk cytogenetics
       * IPSS score of INT-2 or greater
       * Treatment-related MDS
       * MDS diagnosed before age 21 years
       * Progression on or lack of response to standard DNA-methyltransferase inhibitor therapy
       * Life-threatening cytopenias, including those generally requiring greater than weekly transfusions
  7. Interferon- or imatinib-refractory CML in first chronic phase, or non-blast crisis CML beyond first chronic phase
  8. Philadelphia chromosome negative myeloproliferative disease (including myelofibrosis)
  9. Chronic myelomonocytic leukemia
  10. Juvenile myelomonocytic leukemia

      * For patients with SLL, CLL, or prolymphocytic leukemia, < 20% of bone marrow cellularity involved by this process
      * Adequate end-organ function:
* Left ventricular ejection fraction greater than or equal to 35%
* Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST < 5 x ULN
* FEV1 and FVC > 40% of predicted; or in pediatric patients, if unable to perform pulmonary function tests due to young age, oxygen saturation >92% on room air

  * ECOG performance status < 2 or Karnofsky or Lansky score > 60

Exclusion Criteria:

* Pregnant or breast-feeding
* Uncontrolled infection Note: Infection is permitted if there is evidence of response to medication. Eligibility of HIV infected patients will be determined on a case-by-case basis.
* Any previous BMT within 3 months prior to start of conditioning
* Active extra-medullary leukemia or known active Central Nervous System (CNS) involvement by malignancy. Such disease treated into remission is permitted.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Kasamon, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sydney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BMT Allogenic Transplantation: Fludarabine, Busulfan, Cyclophosphamide, Tacrolimus,: Fludarabine 30 mg/m2 IV once a day for 4 days Busulfan 0.8 mg/kg IV every 12 hours for 4 days Cyclophosphamide 50 mg/kg IV daily for 2 days
Period: Overall Study
Arm/Group | BMT Allogenic Transplantation
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 49 [3 to 73]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 2
Sex/Gender, Customized [Number; unit: participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Chimerism in Unsorted Peripheral Blood
Description: Percentage of participants achieving full-donor chimerism in unsorted peripheral blood.
Time Frame: Day 60
Population: The trial has been terminated early since stopping rule criteria were met (high graft failure rate). Data were not analyzed.
Groups:
- BMT Allogenic Transplantation: Reduced-intensity transplant with a fludarabine- and busulfan-based preparative regimen. GVHD prophylaxis with cyclophosphamide, tacrolimus, and mycophenolate mofetil.
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 0

2. Primary Outcome: Chimerism in CD3+ Sorted Peripheral Blood
Description: Percentage of participants achieving full-donor chimerism in CD3+ sorted peripheral blood
Time Frame: Day 60
Population: as for outcome 1
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Percentage of participants alive
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Percentage of participants alive without disease relapse or progression.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Relapse
Description: Percentage of participants experiencing disease relapse or progression
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 0

6. Secondary Outcome: Non-relapse Mortality
Description: Percentage of participants who died due to BMT-related reasons
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | BMT Allogenic Transplantation
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Graft-versus-host-disease (GVHD)
Description: Percentage of participants experiencing acute and chronic GVHD. Acute GVHD is graded by Przepiorka criteria. Chronic GVHD is graded by NIH consensus criteria and Seattle criteria.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Transplant
Number analyzed (Participants) | 0

8. Secondary Outcome: Graft Failure
Description: Percentage of participants who failed to engraft.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant
Number analyzed (Participants) | 15
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 year
Description: Data was collected systematically through at least Day 60 by investigator assessment at protocol-specified visits.
Arm/Group | Transplant
All-Cause Mortality (participants affected / at risk) | 9/15
Serious Adverse Events (participants affected / at risk) | 11/15
Other Adverse Events (participants affected / at risk) | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant (N=15)
Infection (Infections and infestations) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant (N=15)
nausea (Gastrointestinal disorders) | 1 (2)
fever (General disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
hallucinations (Psychiatric disorders) | 1 (1)
Elevated liver enzymes (Investigations) | 1 (1)
Elevated total bilirubin (Investigations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection (Infections and infestations) | 4 (4)
Febrile neutropenia (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes